CLINICAL TRIAL: NCT04748822
Title: Factors Associated With Quality of Life in Patients With Alcohol Use Disorder
Brief Title: Quality of Life in Patients With Alcohol Use Disorder
Acronym: QUALIFACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A02853-36
Record Dates: First submitted 2021-01-19; First posted 2021-02-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Surveys and Questionnaires; Ethanol

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality of life of patients with AUD. (Other): Patients' demographic data, socioeconomic status, physical diseases, medication use, clinical features of AUD, psychiatric variables, impulsivity, autonomy, sexual functioning, sleep quality, and cognitive functioning will be measured at baseline. The Alcohol Quality of Life Scale (AQoLS) will be completed at baseline and at 6-month follow-up. Alcohol status (relapse/abstinence) will be assessed at 6 months.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — The Alcohol Quality of Life Scale (AQoLS) will be completed at baseline and at 6-month follow-up. Alcohol status (relapse/abstinence) will be assessed at 6 months.
  Other Names: Alcohol Quality of Life Scale (AQoLS) and Alcohol status

SUMMARY:
The primary purpose of this study is to investigate the factors associated with quality of life of patients with alcohol use disorder (AUD) undergoing a detoxification program (cross-sectional analysis). The secondary purpose is (1) to identify the factors associated with change in quality of life between baseline and 6-month follow-up, and (2) to identify the factors associated with alcohol relapse at 6 months (longitudinal analyses).

DETAILED DESCRIPTION:
The standard DSM-5-based clinical assessment of AUD includes the number of AUD criteria (between 2 and 11) as well as various parameters related to the patterns of alcohol use (e.g., frequency of use, frequency of heavy use). In the contemporary clinical practice, more "functional" assessment tools are emerging such as quality of life, autonomy, cognitive functioning, but also other non-specific lifestyle habits, such as sleep quality and sexual functioning. These indicators are important because they define the broad impact of AUD on individual's life, and they are part of the overall rehabilitation, beyond the mere question of the relationship to alcohol. However, the determinants of quality of life of patients with AUD patients undergoing a detoxification program, and the factors associated with change in quality of life are not well identified.

This prospective cohort study will recruit 200 patients undergoing a detoxification program (home-based or in addiction services). Patients' demographic data, socioeconomic status, physical diseases, medication use, clinical features of AUD, psychiatric variables, impulsivity, autonomy, sexual functioning, sleep quality, and cognitive functioning will be measured at baseline. The Alcohol Quality of Life Scale (AQoLS) will be completed at baseline and at 6-month follow-up. Alcohol status (relapse/abstinence) will be assessed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 AUD criteria
* At least 18 years of age
* Within the 10th and 21st day of a detoxification program.

Exclusion Criteria:

* Communication difficulties (insufficient level of French, major hearing or visual impairment, major cognitive deficit)
* Under guardianship
* Under justice control
* Cannot be reached by phone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Quality of life in patients with AUD. | Within the 10th and 21st day of the detoxification program (baseline assessment).
  Alcohol Quality of Life Scale.

SECONDARY OUTCOMES:
Quality of life in patients with AUD 6 months after the detoxification program. | 6 months after the baseline assessment.
  Alcohol Quality of Life Scale.
Alcohol status | 6 months after the baseline assessment.
  Alcohol (relapse/abstinence)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, MD, PhD, Principal Investigator — CH LE VINATIER; LOUIS FERDINAND LESPINE, MD, Study Director — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No